CLINICAL TRIAL: NCT03942822
Title: Effect of a Chia Supplemented Diet (Salvia Hispanica) on the Cardiometabolic Risk Profile in Patients With NAFLD (Non Alcoholic Fatty Liver Disease)
Brief Title: Chia Supplementation and Non Alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Aida Medina Urrutia, Medical sience investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-980
Record Dates: First submitted 2019-04-25; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Dietary Modification
Keywords: Non-Alcoholic Fatty Liver Disease; Milled chia seed suplementation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chia supplemented group (Experimental): 8 weeks of 25 g/day of milled chia supplemented-isocaloric diet
  Interventions: Dietary Supplement: Milled chia seeds

INTERVENTIONS:
Dietary Supplement: Milled chia seeds — 8 weeks of an isocaloric diet supplemented with 25 g/day of milled chia

SUMMARY:
Parallel to epidemic obesity, non-alcoholic fatty liver disease (NAFLD) prevalence has markedly increased during the last years, and recent data point out that one of three adults courses with this disease. NAFLD etiopathogeny is multifactorial, an inadequate diet characterized by high fructose content and deficient consumption of omega-3 fatty acids, scarce physical activity, excess abdominal visceral fat (AVF), insulin resistance, and genetic susceptibility have shown to be relevant determinants. Although NAFLD can progress to cirrhosis and hepatic carcinoma, its most frequent complications are type 2 diabetes mellitus (DM2) and coronary artery disease (CAD); therefore, NAFLD is considered a multisystemic disease and a public health problem.

Currently, no specific pharmacological treatment is available for NAFLD, hence, modifications in life style, including weight loss by caloric restriction and increased physical activity, are still the treatment of choice for this type of patients. Recent studies indicate that the supplementation of the diet with omega-3 fatty acids of marine origin (eicosapentanoic acid [EPA]/docosahexaenoic acid [DHA]) and the Mediterranean-style diet (rich in omega-3, antioxidants, and fiber) are efficient for NAFLD treatment, because they diminish the intrahepatic fat content and improve the metabolic profile, even in non-caloric restriction diets. However, the socioeconomic and cultural characteristics make the consumption of these food difficult in some populations, which has led to the search of alternative vegetal sources rich in these nutrients.

Although, there is evidence in animal models suggesting that chia (Salvia hispanica L.) could be an alternative able to reduce the intrahepatic fat content, its effect on NAFLD has not been studied in humans. Hence, the objective of this study was to analyze whether the consumption of an isocaloric diet supplemented with 25 g/day of chia can diminish NAFLD and the metabolic anomalies that accompany the disease.

DETAILED DESCRIPTION:
Participants were chosen from the control group of the Genetics of the Atherosclerotic Disease (GEA, for its initials in Spanish) study, performed at the Institute National of Cardiology "Ignacio Chávez" in Mexico City, Mexico. The protocol was approved by the Research and Ethics Committee of the Instituto Nacional de Cardiología "Ignacio Chavez" under the number 16-980. Candidates that accepted to participate in the study signed voluntarily the informed consent.

In order to know eating habits and standardize macronutrient dietary composition, 24-hour dietary recalls will be applied in the first visit, considering two weekdays and one day of the weekend. Patients will be instructed to maintain constant their physical activity throughout the study. To standardize macronutrient dietary composition, an isocaloric diet (55% carbohydrate, 30% fat, and 15% protein diet) will be indicated two weeks before starting chia supplementation. After this, participants will be instructed to keep up this macronutrient composition during all the intervention period. 30 packages of 25 g of chia seeds will be provided to each patient monthly, with the instruction to mill one package per day, pointing out on the relevance of consume the milled chia accompanied by with water, salads, cereal, or other dishes, from breakfast through lunch but always before 6:00 PM. To favor treatment adherence and record adverse events (loss appetite loss, constipation, diarrhea, flatulence and nausea, allergy or chía chia intolerance), patients will be contacted once a week during the intervention. Adherence will be determined by counting empty chia packages, and evaluation of alpha linolenic acid (ALA) concentration in plasma, which is the chia's seeds main fatty acid compound.

Anthropometric evaluation, laboratory test, and computed tomography studies will be made at baseline and after the 8-wk intervention.

Nutritional intervention and food intake evaluation In order to know eating habits and standardize macronutrient dietary composition, 24-hour dietary recalls will be applied in the first visit, considering two weekdays and one day of the weekend. Patients will be instructed to maintain constant their physical activity throughout the study. To standardize macronutrient dietary composition, an isocaloric diet (55% carbohydrate, 30% fat, and 15% protein diet) will be indicated two weeks before starting chia supplementation. After this, participants will be instructed to keep up this macronutrient composition during all the intervention period. 30 packages of 25 g of chia seeds will be provided to each patient monthly, with the instruction to mill one package per day, pointing out on the relevance of consume the milled chia accompained by with water, salads, cereal, or other dishes, from breakfast through lunch but always before 6:00 PM. To favor treatment adherence and record adverse events (loss appetite loss, constipation, diarrhea, flatulence and nausea, allergy or chía chia intolerance), patients will be contacted once a week during the intervention.

Adherence will be determined by counting empty chia packages, and evaluation of alpha linolenic acid (ALA) concentration in plasma, which is the chia's seeds main fatty acid compound. Participants wre excluded when the adherence was lower tan 80% according to the package counting, or when plasma ALA concentration increased less than 30%.

Anthropometric evaluation, laboratory test, and computed tomography studies will be made at baseline and after the 8-wk of diet intervention.

Anthropometric evaluation: Weight and height will be recorded using a calibrated scale and wall stadiometer, with an accuracy of 0.1 Kg kg and 0.1 cm, after removing excess clothing and shoes. The body mass index (BMI) was calculated as weight (kg)/height (m2). Waist circumference will be measured with a non-stretch tape, at the midway between the lowest rib and the iliac crest without clothes around the waist.

Laboratory tests: After 10-h fasting and 20 min in sitting position, venous blood will be collected in assay tubes without anticoagulant and in tubes with K2-EDTA (1.8 mg/mL). Glucose, total cholesterol, triglyceride, and high density lipoprotein cholesterol (HDL-C) concentrations will be determined using direct standard enzymatic colorimetric methods on a COBAS c311 (Roche Diagnostics, Mannheim, Germany). Low density lipoprotein cholesterol (LDL-C) concentration was estimated using the De Long formula. The reproducibility and precision of these determinations in our laboratory is assessed by the Center for Disease Control and Prevention Lipids Standardization Program (LSP-CDC, Atlanta, GA, USA). Plasma free fatty acids (FFA) will be measured by an enzymatic-colorimetric assay (Wako Diagnostics, Chuo-Ku Osaka, Japan). Total fatty acids, including ALA will be extracted according to Folch method, and analyzed in a Shimadzu GC-8A gas chromatograph equipped with an SP2330 capilar column (25m x 0.25 mm x 0.25). Fatty-acid concentrations will be calculated in relation to heptadecanoic acid methyl ester as internal standard, fatty acids peaks will be identified by using the Supelco 37 component FAME Mix (CRM47885). A plasma control sample will be run in each extraction assay, to obtain an ALA inter-assay coefficient variation.

Computed tomography study: Computed tomography (CT) is a validated method for measuring visceral adipose tissue (VAT) and evaluate non alcoholic fatty liver disease. In the present study, these measurements will be obtained using a 64-slice scanner (Somatom Cardiac Sensation 64, Forcheim, Bavaria, Germany). To determine the liver and spleen attenuation index, a single slice CT scan is obtained at the level of T11-T12 or T12-L1. Fatty liver is defined as a liver/spleen attenuation ratio lower than 1.0. To calculate the amount of total abdominal tissue (TAT) and VAT, a single slice scan is obtained at the level of L4-L5, the area is expressed in square centimeters (cm2). Subcutaneous abdominal tissue (SAT) was calculated by subtracting the VAT from the TAT area.

ELIGIBILITY:
Inclusion Criteria:

* Tomographic diagnosis of NAFLD
* Insulin resistance (HOMA-IR > 3.7 in women and 3.4 in men)

Exclusion Criteria:

* Previous diabetes diagnosis
* Use of hypoglycemic or hypolipidemic medications
* Significant weight changes during the previous 3 months (± 5% of their habitual weight)
* Consumption of vitamins, herbal or food supplements
* Gastrointestinal, renal, or hepatic diseases
* Eating, psychiatric or cognitive disorders that would hinder them of understanding and complying with the instructions of the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Effect of a chia (Salvia hispanica L.) supplemented diet in patients with non-alcoholic fatty liver | 8 weeks
  To assess the effect of 25 g/day of milled chia in 25 patients with NAFLD.Improvement of LSAI (liver spleen attenuation index) measured by computed tomography In a single-arm experimental design study
Effect of chia on plasma levels of alpha linolenic acid | 8 weeks
  Increase in Alpha linolenic acid with chia supplemented diet. Measured by gas chromatography.

SECONDARY OUTCOMES:
Effect of chia on lipid parameters | 8 weeks
  Improvement of lipid parameters (total colesterol, LDL-C, triglycerides, HDL-C) including free fatty acids

REFERENCES:
- [Derived] Medina-Urrutia A, Lopez-Uribe AR, El Hafidi M, Gonzalez-Salazar MDC, Posadas-Sanchez R, Jorge-Galarza E, Del Valle-Mondragon L, Juarez-Rojas JG. Chia (Salvia hispanica)-supplemented diet ameliorates non-alcoholic fatty liver disease and its metabolic abnormalities in humans. Lipids Health Dis. 2020 May 19;19(1):96. doi: 10.1186/s12944-020-01283-x. PMID 32430018